CLINICAL TRIAL: NCT01648465
Title: Phase II Multicenter Single-arm Study Evaluating the Safety and Efficacy of Everolimus as a First-line Treatment in Newly-diagnosed Patients With Advanced GI Neuroendocrine Tumors.
Brief Title: Study of Everolimus Treatment in Newly-diagnosed Patients With Advanced Gastrointestinal Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE 67/12; 2011-006160-48 (EudraCT Number)
Record Dates: First submitted 2012-07-13; First posted 2012-07-24 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Gastrointestinal Tumors; Pancreatic Tumors; Gastrointestinal Neuroendocrine Tumors; Pancreatic Neuroendocrine Tumors
Keywords: metastatic; unresectable; well or moderately differentiated; advanced
MeSH Terms: conditions — Digestive System Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus 10mg(2x5mg)orally once daily until disease progression, unacceptable toxicity or consent withdrawal
  Other Names: Afinitor; RAD001

SUMMARY:
The purpose of this study is to explore the efficacy and safety of everolimus administered as a first-line treatment in newly-diagnosed patients with advanced or inoperable Gastrointestinal (GI) or pancreatic neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years of age.
2. Newly diagnosed patients with biopsy-proven well or moderately differentiated advanced (metastatic or unresectable) GI or pancreatic neuroendocrine tumor.
3. Measurable disease based on RΕCIST 1.1 using a triphase CT scan or multi-phase MRI scan.
4. Patients with a ki-67 measurement <20% prior to their enrollment to the study.
5. Performance status 0-2 on the WHO scale.
6. Adequate bone marrow function as shown by:ANC ≥ 1.5 x 10^9/L,Platelets ≥ 100 x 10^9/L,Hemoglobin > 9 g/dL.
7. Adequate liver function as shown by:Serum bilirubin ≤ 1.5 x ULN,ALT/SGPT and AST/SGOT ≤ 2.5 x ULN (ή ≤ 5 x ULN in patients with known liver metastases),INR < 1.3 (INR < 3 in patients treated with anticoagulants).
8. Adequate renal function as shown by: serum creatinine ≤ 1.5 x ULN.
9. Fasting serum cholesterol ≤ 300 mg/dL or ≤ 7.75 mmol/L and fasting triglycerides ≤ 2.5 x ULN. Note: In case one or both the above upper limits are exceeded, patient enrollment can only be performed upon proper antilipidemic treatment initiation.
10. Women of childbearing potential, with a negative serum or urine pregnancy test within 48 hours prior to first study treatment administration.
11. Signed informed consent form obtained before any trial related activity, including the screening phase, according to the applicable law and ICH/GCP requirements.
12. Signed informed consent for the use of biological and genetic material

Exclusion Criteria:

1. Patients with poorly differentiated or undifferentiated GI or pancreatic neuroendocrine carcinoma.
2. Previous or concurrent cytotoxic chemotherapy, immunotherapy or radiotherapy.
3. Hepatic artery embolization or cryoablation of hepatic metastasis within 1 month of study enrollment.
4. Prior therapy with mTOR inhibitors (for example sirolimus, temsirolimus, everolimus).
5. Patients receiving chronic treatment with corticosteroid immunosuppressives.
6. Uncontrolled diabetes mellitus as defined by fasting serum glucose > 1.5 x ULN.
7. Patients who have any severe and/or uncontrolled medical conditions such as:

   * unstable angina pectoris, symptomatic congestive heart failure NYHA class II, III, IV, myocardial infarction ≤ 6 months prior to enrollment, serious uncontrolled cardiac arrhythmia (LVEF < 50 %)
   * active or uncontrolled severe infection
   * cirrhosis, chronic active hepatitis, chronic persistent hepatitis or inadequate hepatic function (ALT/SGPT and AST/SGOT > 5 x ULN)
   * inadequate bone marrow (ANC < 1.5 x 10^9/L, platelets < 100 x 10^9/L, hemoglobin ≤ 9 g/dL) or renal failure (serum creatinine > 1.5 x ULN
   * severely impaired lung function (patients needing oxygen support).
8. Active bleeding diathesis or on oral treatment with vitamin K antagonists (apart from low-dose coumadine).
9. Performance status ≥ 3 on the WHO scale.
10. Patients with a known history of HIV seropositivity. Screening for HIV infection at baseline is not required.
11. No other prior or concurrent malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, or treated in situ cancer of the cervix, or any other cancer from which the patient has been disease free for ≥ 3 years.
12. Patients within 28 days post-major surgery (e.g. intra-thoracic, intrabdominal or intra-pelvic), open biopsy, or significant traumatic injury to avoid wound healing complications. Minor procedures and percutaneous biopsies or placement of vascular access device require 7 days prior to study entry. Note: Patients must have recovered from the acute effects of surgery prior to enrollment.
13. Female patients who are pregnant or nursing (lactating).
14. Adults with reproductive potential who are not using effective birth control methods. If barrier contraceptive measures are being used, these must be continued throughout the study by both sexes.
15. Patients participating in another clinical trial or receiving an investigational drug.
16. Patients unwilling or unable to comply with the protocol at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
15 month PFS (Progression-Free Survival) rate | 15 months
  To determine the rate of PFS patients at 15 months of treatment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Defined as the time from the date of enrollment to the date of 1st radiologically documented disease progression or disease related death,assessed up to 36 months.
Overall Survival (OS) | Defined as the time from the date of enrollment to the date of death from any cause,assessed up to 36 months.
Evaluation of best response to treatment and the time to best response achievement | Defined as the period from the date of treatment initiation to best response observation date througout the study, assessed up to 15 months.
Assessment of safety | Assessment of adverse events will be performed every 28 days (per cycle) during treatment, assessed up to 16 months.
Association of biologic markers with disease progression | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Koumarianou, Dr, Study Chair — 4th Dept of Internal Medicine, University Hospital "Attikon"
Locations (12):
- Greece (12):
  - 2nd Dept of Internal Medicine, Agios Savvas Cancer Hospital, Athens
  - Dept of Medical Oncology, 251 General Airforce Hospital, Athens
  - 2nd Dept of Internal Medicine, General Hospital of Athens "Hippokratio", Athens
  - 2nd Dept of Internal Medicine, Propaedeutic, University Hospital "Attikon", Athens
  - 4th Dept of Internal Medicine, University Hospital "Attiko", Athens
  - 3rd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens
  - 2nd Dept of Medical Oncology, Metropolitan Hospital, Athens
  - Dept of Medical Oncology, University Hospital of Heraklion, Heraklion
  - Dept of Medical Oncology, Ioannina University Hospital, Ioannina
  - Division of Oncology, Dept of Internal Medicine, University Hospital of Patras, Pátrai
  - Dept of Medical Oncology, Papageorgiou General Hospital, Thessaloniki
  - Dept of Medical Oncology, Thermi Clinic, Thessaloniki

REFERENCES:
- [Derived] Koumarianou A, Pectasides D, Koliou GA, Dionysopoulos D, Kolomodi D, Poulios C, Skondra M, Sgouros J, Pentheroudakis G, Kaltsas G, Fountzilas G. Efficacy and Safety of First-Line Everolimus Therapy Alone or in Combination with Octreotide in Gastroenteropancreatic Neuroendocrine Tumors. A Hellenic Cooperative Oncology Group (HeCOG) Study. Biology (Basel). 2020 Mar 9;9(3):51. doi: 10.3390/biology9030051. PMID 32182791